CLINICAL TRIAL: NCT06995794
Title: Effect Of Kinesio Tape Versus Knee Strap on Osgood Schlatter Disease in Athletic Children
Brief Title: Osgood-Schlatter Disease in Athletic Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, ahmed hosny ibrahim eldersy, physiotherapist, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Osgood-Schlatter disease
Record Dates: First submitted 2025-03-30; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Osgood-Schlatter Disease
MeSH Terms: conditions — Osteochondrosis | interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- effect of Kinesio tape application in Osgood Schlatter disease (Active Comparator): will recieve kinesio tape in addition to traditional exercises program including ultrasoud therapy and heat application.
  Interventions: Other: kinesio tape
- effect of knee strap application in Osgood Schlatter disease (Active Comparator): knee strap in addition to traditional exercises program including ultrasoud therapy and heat application.
  Interventions: Other: knee strap

INTERVENTIONS:
Other: kinesio tape — Kinesio tape a therapeutic tape that's applied strategically to the body to provide lessen pain, reduce swelling, improve performance.
  Arms: effect of Kinesio tape application in Osgood Schlatter disease
Other: knee strap — knee strap is used to support the tibial tuberosity which lessen the pain and enhance performance of the knee
  Arms: effect of knee strap application in Osgood Schlatter disease

SUMMARY:
This study will be conducted to evaluate the effect of using Kinesio tape versus strapping the knee on pain management

DETAILED DESCRIPTION:
Osgood-Schlatter disease is a traction apophysitis of the tibial tuberosity caused by the repetitive pull of the patellar tendon on the tibia. This condition was described separately and simultaneously by Robert Osgood and Carl Schlatter in 1903 as a lesion where the tibial tubercle separates due to repetitive strain by the patellar tendon and becomes tender. Kicking, jumping, sprinting sports, a history of previous Sever's disease, and lower limb muscle tightness are among the risk factors that have been associated with Osgood-Schlatter disease. It is one of the leading causes of anterior knee pain in children and adolescents. Usually, patient history and physical examination are sufficient for diagnosis. It can be easily recognized by local pain, swelling, and tenderness on the tuberosity in one or both knees.

Osgood-Schlatter disease (OSD) is a common pediatric disorder. It is a growth- and sports-associated knee injury with pain around the tibial tuberosity and morphological alterations around the apophysis during adolescent growth. It often results from acute or chronic overload during sports activity, causing inflammation of the patellar tendon insertion on the tibial tuberosity. It was first described in 1903 independently by Osgood in the US and by Schlatter in Switzerland. Classically, the clinical presentation is associated with an insidious onset (usually atraumatic) of anterior functional knee pain over the tibial tuberosity along with a bony prominence, as well as tenderness at the patellar tendon insertion site.

Osgood-Schlatter disease occurs during the apophyseal phase between the ages of 12 and 15 in boys and 8 and 12 in girls. During the maturation phase, the cartilage cells of the proximal part of the tuberosity migrate distally, replacing the fibrocartilage in the middle part. This makes the tuberosity unable to withstand the force exerted by the quadriceps, resulting in micro-avulsions, with secondary ossification. These bone fragments are secondarily incorporated into the remainder of the tibial tuberosity, which can result in sequelae of an enlarged tuberosity. In rare cases, the fragments are not incorporated, and intratendinous bone fragments can remain after growth stops, requiring surgical removal. The pain usually occurs during and after physical activity and might be associated with local swelling. Many patients are completely asymptomatic, with less than 25% reporting pain at the tibial tuberosity apophysis. The age of onset is between 8 and 15 years. Boys experience it more often than girls, with a male-to-female ratio of 3:1. The prevalence of OSD is 9.8%, and it can be bilateral in 20-30% of patients. Many risk factors and activities have been associated with an increased incidence of the pathology.

Treatment is generally conservative, with rest, ice, and specific exercises recommended. It involves limiting activity until inflammation resolves and performing exercises that strengthen the surrounding musculature to reduce stress across the tibial tuberosity. Treatment with the PRICE protocol (Protection, Rest, Ice, Compression, Elevation), physical therapy, and strict activity modification is initiated. Surgical removal of ossicles may be considered. A knee strap can immobilize and protect joints, reduce pain, decrease swelling, and facilitate healing of acute injuries. Knee straps are also used for injury prevention and chronic pain reduction. Infrapatellar strapping is a treatment technique employed for various knee pathologies; however, its effect on pain and functional performance among young athletes has not been studied.

Kinesio Taping is effective in improving pain and joint function in patients with knee osteoarthritis. Kinesiology tape is used in the treatment of muscle, fascia, and tendon symptoms and for performance enhancement by way of continuous receptor stimulation. The natural healing process is instantly enhanced due to improved circulation in the taped area. When a muscle is inflamed, swollen, or stiff, the space between the skin and the muscle is compressed, resulting in constriction and congestion of lymphatic fluid and blood circulation. This compression applies pressure to pain receptors located in the space between the skin and the muscle, relaying discomfort signals to the brain and causing the sensation of pain. Stretching the skin of the affected area before applying Kinesiology Tape ensures that the taped area will form wrinkles when the applied area returns to its neutral position. This wrinkling effect is essential because the lifting of the skin creates more space for lymph and blood flow. Consequently, lymph drainage and blood circulation in the affected area are improved effectively through taping application. The friction between the tissues beneath the skin decreases due to the promoted movement of lymphatic fluid and blood circulation. Pain is reduced as the pressure on the pain receptors lessens. The end result is believed to be reduced muscle fatigue, an increased range of motion, and improved quality of muscle contraction.

ELIGIBILITY:
Inclusion Criteria:

* Children will be included in the study if they fulfil the following criteria:

  1. A medical diagnosis with Osgood Schlatter disease was made by paediatricians or paediatric orthopaedist.
  2. Number of the participate children will be 38 children.
  3. Age ranges from 9 to 15 years.

Exclusion Criteria:

* Children will be excluded from the study if:

  1. They had a permanent deformity (bony or soft tissue contractures).
  2. Children have visual or auditory defects.
  3. Children with intelligence quotient less than 70.
  4. Children who had undergone a previous surgical intervention to knee joint.
  5. A history of epileptic seizure and any diagnosed cardiac or orthopaedic disability that may prevent the use of assessment methods.
  6. Children who are absent in two sessions.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of the effect of knee strap with the effect of Kinesio tape on pain management in Osgood Schlatter disease | baseline
  Pain assessment using visual analogue scale. it is widely used to assess pain using straight horizontal line with a fixed length usually 100mm, the two ends of the line represent the extreme limits of the parameter being measured, the left end represents the worst condition while the right end represent the best condition. zero to ten from left to right, zero means no pain and ten is the worest pain

SECONDARY OUTCOMES:
Range of motion assessment | baseline
  Range of motion using electrical goniometer. Universal goniometer in clinical evaluations of patients (as they are easy to be employed) and electro goniometer in laboratory studies (as they are more accurate) are reliable to test the knee range of motion.
muscle power assessment | baseline
  Muscle strength in the quadriceps may be weaker due to limited exercise, as pain persists. The Lafayette Manual Muscle Tester is used to measure maximal isometric knee extension and flexion. A higher value indicates greater muscle strength
functional assessment | baseline
  Single leg triple hops Functional scale to evaluate the activity pre and post treatment for both groups

CONTACTS AND LOCATIONS:
Overall Officials: samar t elbanna, Study Chair — Kafr Elshekh university

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Greenberg EM, Dyke J, Leung A, Karl M, Lawrence JT, Ganley T. Uninjured Youth Athlete Performance on Single-Leg Hop Testing: How Many Can Achieve Recommended Return-to-Sport Criterion? Sports Health. 2020 Nov/Dec;12(6):552-558. doi: 10.1177/1941738120911662. Epub 2020 May 11. PMID 32392085
- [Background] Shamsi M, Mirzaei M, Khabiri SS. Universal goniometer and electro-goniometer intra-examiner reliability in measuring the knee range of motion during active knee extension test in patients with chronic low back pain with short hamstring muscle. BMC Sports Sci Med Rehabil. 2019 Mar 22;11:4. doi: 10.1186/s13102-019-0116-x. eCollection 2019. PMID 30949343
- [Background] Knapik JJ, Wright JE, Mawdsley RH, Braun JM. Isokinetic, isometric and isotonic strength relationships. Arch Phys Med Rehabil. 1983 Feb;64(2):77-80. PMID 6824423
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Lu Z, Li X, Chen R, Guo C. Kinesio taping improves pain and function in patients with knee osteoarthritis: A meta-analysis of randomized controlled trials. Int J Surg. 2018 Nov;59:27-35. doi: 10.1016/j.ijsu.2018.09.015. Epub 2018 Sep 28. PMID 30273684
- [Background] Davis J, Doyle B, Ishii H, Jayanthi N. S.P.O.R.R.T.-A Comprehensive Approach to the Assessment and Non-Operative Management of Overuse Knee Conditions in Youth Athletes. Curr Rev Musculoskelet Med. 2023 Dec;16(12):627-638. doi: 10.1007/s12178-023-09874-8. Epub 2023 Nov 24. PMID 37999828
- [Background] van Leeuwen GJ, de Schepper EI, Rathleff MS, Bindels PJ, Bierma-Zeinstra SM, van Middelkoop M. Incidence and management of Osgood-Schlatter disease in general practice: retrospective cohort study. Br J Gen Pract. 2022 Mar 31;72(717):e301-e306. doi: 10.3399/BJGP.2021.0386. Print 2022 Apr. PMID 34990396
- [Background] Launay F. Sports-related overuse injuries in children. Orthop Traumatol Surg Res. 2015 Feb;101(1 Suppl):S139-47. doi: 10.1016/j.otsr.2014.06.030. Epub 2014 Dec 30. PMID 25555804
- [Background] Dar G, Mei-Dan E. Immediate effect of infrapatellar strap on pain and jump height in patellar tendinopathy among young athletes. Prosthet Orthot Int. 2019 Feb;43(1):21-27. doi: 10.1177/0309364618791619. Epub 2018 Aug 13. PMID 30101673
- [Background] Logan CA, Bhashyam AR, Tisosky AJ, Haber DB, Jorgensen A, Roy A, Provencher MT. Systematic Review of the Effect of Taping Techniques on Patellofemoral Pain Syndrome. Sports Health. 2017 Sep/Oct;9(5):456-461. doi: 10.1177/1941738117710938. Epub 2017 Jun 15. PMID 28617653
- [Background] Lucenti L, Sapienza M, Caldaci A, Cristo C, Testa G, Pavone V. The Etiology and Risk Factors of Osgood-Schlatter Disease: A Systematic Review. Children (Basel). 2022 Jun 2;9(6):826. doi: 10.3390/children9060826. PMID 35740763
- [Background] Corbi F, Matas S, Alvarez-Herms J, Sitko S, Baiget E, Reverter-Masia J, Lopez-Laval I. Osgood-Schlatter Disease: Appearance, Diagnosis and Treatment: A Narrative Review. Healthcare (Basel). 2022 May 30;10(6):1011. doi: 10.3390/healthcare10061011. PMID 35742062
- [Background] Lyng KD, Rathleff MS, Dean BJF, Kluzek S, Holden S. Current management strategies in Osgood Schlatter: A cross-sectional mixed-method study. Scand J Med Sci Sports. 2020 Oct;30(10):1985-1991. doi: 10.1111/sms.13751. Epub 2020 Aug 26. PMID 32562293
- [Background] Bezuglov EN, Tikhonova capital A, Cyrilliccapital A, Cyrillic, Chubarovskiy PV, Repetyuk capital A, CyrillicD, Khaitin VY, Lazarev AM, Usmanova EM. Conservative treatment of Osgood-Schlatter disease among young professional soccer players. Int Orthop. 2020 Sep;44(9):1737-1743. doi: 10.1007/s00264-020-04572-3. Epub 2020 Apr 28. PMID 32346752
- [Background] Neuhaus C, Appenzeller-Herzog C, Faude O. A systematic review on conservative treatment options for OSGOOD-Schlatter disease. Phys Ther Sport. 2021 May;49:178-187. doi: 10.1016/j.ptsp.2021.03.002. Epub 2021 Mar 9. PMID 33744766
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/

DOCUMENTS (2):
  • Study Protocol (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT06995794/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT06995794/SAP_001.pdf